CLINICAL TRIAL: NCT05653804
Title: Impact of Tele-visit Versus Home Visit by Home Care Provider on Compliance With Continuous Positive Airway Pressure (CPAP) Therapy of Patients With Obstructive Sleep Apnea Syndrome
Brief Title: Impact of Tele-visit on Patients Continous Positive Airway Pressure (CPAP) Follow-up by Home Care Provider
Acronym: i-tech PPC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AGIR à Dom (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022-A02309-34
Record Dates: First submitted 2022-11-18; First posted 2022-12-16 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Obstructive Sleep Apnea
Keywords: tele-visit
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: Prospective, interventional, randomized controlled, open-label, single-center, multi-site
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tele-visit by HCP (Experimental): Patients receive a annual CPAP remote visit by HCP technician, then home visit the following year
  Interventions: Procedure: tele-visit
- home visit by HCP (No Intervention): Standard care : patients receive an annual CPAP home visit by HCP technician

INTERVENTIONS:
Procedure: tele-visit — The remote visit content for CPAP follow up is based on home visit framework and carried out from a secure platform for sharing health data.
  Arms: tele-visit by HCP

SUMMARY:
To determine the impact of telecare on continous positive airway pressure (CPAP) patients follow up by home care provider (HCP)

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) syndrome is a chronic respiratory pathology affecting 4% of french adult population and reference treatment for moderate to severe forms of obstructive sleep apnea syndrome (OSA) is continuous positive airway pressure (CPAP).

However, CPAP treatment is binding, so nearly a quarter of patients abandoning treatment at 1 year and nearly half of them at 3 years. Support for these patients on CPAP must therefore be optimal and seek patient satisfaction; HCP (Home Care Provider) plays an important role in this follow-up.

Since 2018 in France, teleconsultation entered on common law but was little used. The pandemic has disrupted the habits of care and patients monitoring by developing remote monitoring. Home Care Providers (HCP) have also been forced to organize remote monitoring, particularly for the annual follow-up visit (technical tele-visit).

The impact of the annual follow-up visits of HCP by tele-visit has never been clinically evaluated. If its clinical relevance were demonstrated and patient satisfaction confirmed, this follow-up modality could become, like telecare, a new standard for the follow-up of patients on CPAP.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* CPAP ≥ 12 months and annual followed by "AGIR à dom" health care provider.
* Compliance with CPAP ≥ 4h/night and AHI ≤ 5 events/hour on machine report for the 3 months prior to inclusion

Exclusion Criteria:

* Follow-up by AGIR à dom. for an other service than package F9.1 : CPAP follow-up and remote monitoring
* Unacceptable level of mask leakage
* Patient unavailable or willing to move within the next 12 months to an area not covered by AGIR à dom.
* Patient considered by the investigator to be unfit for a tele-visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2026-05-11 (Estimated); Study Completion 2027-05-11 (Estimated)

PRIMARY OUTCOMES:
To compare CPAP compliance between the two management modalities | Over the 3 months (tele)visit follow-up
  CPAP mean compliance between intervention and control groups, adjusted for the three months prior to inclusion : in hours/day, collected on the CPAP remote monitoring report

SECONDARY OUTCOMES:
To compare overall patient satisfaction between the two management modalities | Immediately after the (tele-)visit follow-up
  The Consumer Satisfaction Questionnaire (CSQ-8) mean score between intervention and control groups, after the CPAP (tele-)visit follow-up .
  The overall score is calculated by adding the respondent's evaluation score (item evaluation) for each item on the scale. For the CSQ-8 version, the scores therefore range from 8 to 32, with higher values indicating greater satisfaction.
To compare the impact on daytime sleepiness between the two management modalities | At 3 months after (tele-)visit follow-up
  Epworth Sleepiness Scale (ESS) mean score between intervention and control group.
  All items are assumed to be integers (0-3). The ESS score is the sum of 8 item scores.
  0-10 = normal range of sleepiness in healthy adults 11 to 14 = mild sleepiness 15 to 17 = moderate sleepiness 18 to 24 = severe sleepiness
To compare impact on quality of life between the two management modalities | At 3 months after (tele-)visit follow-up
  The EuroQol 5 Dimensions - 5 levels (EQ5D-5L) questionnaire mean score between intervention and control group, adjusted on the baseline score.
  it's composed of two parts : A visual analog scale (20 cm line, graduated from 0 to 100 where patient indicates his or her current state of health, 0 being the worst and 100 the best)
  the completion of 5 items evaluating mobility, autonomy, daily activities, pain or discomfort and anxiety or depression.
  1. indicating no problem
  2. indicating slight problems
  3. indicating moderate problems
  4. indicating severe problems
  5. indicating unable to/extreme problems Each state is referred to by a 5-digit code.
To compare CPAP compliance in medium term between the two management modalities | Over the 12 months (tele)visit follow-up
  CPAP mean compliance between intervention and control group : in hours/day, collected on the CPAP remote monitoring report
To compare impact on CPAP continuation between the two management modalities | Over the 12 months (tele)visit follow-up
  Rate of CPAP removal between intervention and control group ; the number of CPAP unbundling among participants
To compare treatment effectiveness between the two management modalities | Over the 12 months (tele)visit follow-up
  Apnea Hypopnea Index (AHI) mean between intervention and control group. AHI corresponds to the number of apneas and hypopneas per hour of sleep, collected on the CPAP remote monitoring report.
To compare treatment quality on mask leakage between the two management modalities | Over the 3 months (tele)visit follow-up
  Leakage mean level between intervention and control group
To compare occurrence frequency of CPAP-related adverse effect(s) between the two management modalities | Over the 3 months (tele)visit follow-up
  The Side-Effects to CPAP treatment Inventory (SECI) mean score between the intervention and control group.
  Each of the 15 items relating to side effects associated with CPAP treatment has three subscales: frequency, breadth of the side effect, and impact on CPAP use.
  For each subscale, the patient will complete a five-point Likert-type scale, so the possible range for each subscale is 15 to 75.
  A higher score indicates greater frequency of side effects, greater breadth of side effects, and greater intensity of side effects.
To compare follow-up impact in addition to the annual visit between the two management modalities | Over the 12 months (tele)visit follow-up
  Mean number of calls and visits made per patient between control and intervention group
To evaluate failed visits number between the two care modalities | Over the 12 months (tele)visit follow-up
  Mean number of (tele-)visits requiring a reprogramming (absence, technical problem, last minute deprogramming, home visit...)
To evaluate patient satisfaction with tele-visits | Immediately after the (tele-)visit follow-up
  The Televisit Satisfaction Questionnaire (TSQ) mean score
  14 items, rated between 1 and 5 by the patient. The sum of the items corresponds to a score ranging from 14 to 70.
To evaluate technician satisfaction with tele-visits | Immediately after the (tele-)visit follow-up
  The Televisit Satisfaction Questionnaire (TSQ) questionnaire mean score
  14 items, rated between 1 and 5 by the patient. The sum of the items corresponds to a score ranging from 14 to 70.
Comparison of the environmental impact associated with the two patient follow-up methods (home visit versus tele-visit) | Over the 12 months (tele)visit follow-up
  Comparison of the carbon emissions generated by each care modality, calculated over the entire patient participation period and expressed in kgCO₂e, considering only the impact of the follow-up method itself, without including the individual use of the CPAP device.

OTHER OUTCOMES:
To evaluate patient overall satisfaction regarding clinical study participation | Over the 3 months (tele)visit follow-up
  Survey Satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Jean Christian BOREL, PhD, Principal Investigator — AGIR à Dom
Locations (1):
- AGIR à dom., Meylan, France